CLINICAL TRIAL: NCT02156856
Title: Stroke Volume Analysis During Aortic Valve Replacement Trial
Acronym: standart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Sander, Univ.-Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA1/060/13
Record Dates: First submitted 2014-05-20; First posted 2014-06-05 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Hemodynamic Monitoring; Cardiac Output; Cardiac Surgery
Keywords: hemodynamic monitoring; cardiac output; cardiac surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodynamic optimisation
- No hemodynamic optimisation

SUMMARY:
Compromised peripheral tissue oxygenation during surgery may lead to worse patient outcome, mainly due to post-operative infections or heart failure. Insufficient stroke volume and/or cardiac output due to hypovolemia or cardiac defects play a central role in causing poor peripheral tissue oxygenation. In order to assess stroke volume, there are numerous invasive and non-invasive methods available. Up to the present date it is unknown, if these methods may by used interchangeably in patients with severe cardiac defects like aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* scheduled transcatheter aortic valve implantation
* signed patient consent form
* aged 18 or older by time of surgery
* no participation in other clinical trials

Exclusion Criteria:

* pregnant or breast-feeding women
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery at a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of stroke volume (ml) before TAVI (transcatheter aortic valve implantation) by means of (1) FloTrac, (2) transesophageal doppler echocardiography, (3) pulmonary thermodilution via pulmonary artery catheter | Before Surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Measurement of cardiac output (l/min) before TAVI (transcatheter aortic valve implantation) by means of (1) FloTrac, (2) transesophageal doppler echocardiography, (3) pulmonary thermodilution via pulmonary artery catheter | Before Surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Measurement of stroke volume (ml) after TAVI (transcatheter aortic valve implantation) by means of (1) FloTrac, (2) transesophageal doppler echocardiography and (3) pulmonary thermodilution via pulmonary artery catheter | After surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Accordance of stroke volume and cardiac output measurements assessed by (1) FloTrac, (2) transesophageal doppler echocardiography and (3) pulmonary thermodilution via pulmonary artery catheter AFTER ADMINISTRATION OF FLUID BOLUS | Before and after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Accordance of stroke volume and cardiac output measurements assessed by two of the mentioned methods [i.e. (1) FloTrac, (2) transesophageal doppler echocardiography and (3) pulmonary thermodilution via pulmonary artery catheter] | Before and after Surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Measurement of cardiac output (l/min) after TAVI (transcatheter aortic valve implantation) by means of (1) FloTrac, (2) transesophageal doppler echocardiography and (3) pulmonary thermodilution via pulmonary artery catheter | After Surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks

OTHER OUTCOMES:
oxygen delivery (ml) | Before and after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
image quality of echocardiography | Before and after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Length of stay on ICU | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Cumulative rate of infections | after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
incidence of delirium after surgery | after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
dosage of inotropic medication (mg/d) | after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
length of hospital stay | after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks
incidence of stroke | after surgery; participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berin, Berlin, State of Berlin, Germany